CLINICAL TRIAL: NCT06327906
Title: A Series of Studies Based on a Prospective Birth Cohort of Infants With Allergy and Neurodevelopmental Disorders in China
Brief Title: A Prospective Birth Cohort of Infants With Allergy and Neurodevelopmental Disorders in China
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: qilu000002
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-10

CONDITIONS: Child Allergy; Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dry blood spots were collected and cryopreserved at -80 °C for gene sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, a birth cohort was established to demonstrate the causal relationship between allergies and neurodevelopment disorders in infants and young children, and to find out the influencing factors of neurodevelopment disorders in early life.

DETAILED DESCRIPTION:
In this study, a birth cohort was established, and infants were divided into two groups according to inclusion and exclusion criteria ( see study design ). One group was allergic group, and the other group was control group. The two groups will be followed up for up to 6 years, and specimens ( blood, urine, feces ) and test data ( height, weight, GESELL, etc. ) will be retained during the follow-up period. The outcome indicators were ASD, ADHD or LD, and DSM-5 was used as the diagnostic criteria.

ELIGIBILITY:
Inclusion Criteria:

* ①Allergic questionnaire results were positive.

  * The living area is Jinan City and its surrounding areas in Shandong Province, which is convenient for follow-up.

Exclusion Criteria:

* There is a clear diagnosis of brain developmental disorders

  * Psychological diseases

    * History of craniocerebral trauma or brain organic disease ④Major physical diseases ⑤Visual and auditory disorders ⑥ Epilepsy ⑦Intellectual disabilities

Ages: 1 Minute to 42 Days | Sex: All
Age Groups: Child
Study Population: The obstetrics department of Qilu Hospital of Shandong University recruit pregnant women. After the delivery of pregnant women, the newborns will included in the cohort.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
ASD | from 2023-11-15 to 2026-11-15
  with diagnostic criteria of DSM-V ASD, and ADOS, CARS auxiliary diagnosis.
ADHD | from 2023-11-15 to 2029-11-15
  with diagnostic criteria of DSM-V ADHD, and SNAP-Ⅳ, CONNER auxiliary diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: cao aihua, post-doctoral, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No